CLINICAL TRIAL: NCT04725500
Title: Engineering Evaluation of the Vector NIV Device in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Vector Engineering Clinical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRC-HRC-VectorENG -2018-10241
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: COPD
Keywords: Non Invasive Ventilation; Expiratory Flow Limitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Auto-titrating EPAP (Experimental): ExpiraFlowTM technology- Non-invasive ventilator that auto titrates EPAP to abolish Expiratory flow limitation.
  Interventions: Device: Auto-Titrating EPAP

INTERVENTIONS:
Device: Auto-Titrating EPAP — In the Auto-titrating EPAP mode, the device automatically adjusted EPAP to the minimum level able to abolish tidal expiratory flow limitation.

SUMMARY:
This study aimed to validate a novel automatic non-invasive ventilation (NIV) mode that continuously adjusts expiratory positive airway pressure (EPAP) to the lowest value that abolishes tidal expiratory flow limitation (EFL). The investigator conducted a prospective, non-randomized, study on stable chronic obstructive pulmonary disease (COPD) patients that may or may not be treated currently with NIV. Patients were studied in a sleep lab on a single night with the auto - titrating EPAP that adjusts to abolish tidal EFL. The primary endpoint was to evaluate the behavior of the EPAP during the night. Additionally, a sub-group of patients used the device at home for a 2 week period. EPAP behavior was assessed during this 2 week period.

DETAILED DESCRIPTION:
Tidal Expiratory Flow Limitation (EFLT) is the inability to increase expiratory flow despite increasing effort. Especially in patients with mild to severe COPD, EFL can present challenges when receiving mechanical ventilation. To overcome EFLT expiratory positive airway pressure (EPAP) is applied; however, a single level or fixed EPAP may not overcome the airflow obstruction. The current study was undertaken to explore the variability of EFLT determined using Forced Oscillation Technique (FOT) to dynamically measure lung reactance (∆Xrs) and to evaluate the ability of automatically adjusted EPAP (PEEPopt) to over come EFLT overnight and over a two week period.

In this prospective non-randomized trial, an unreleased noninvasive ventilator set in an S/T mode applied continuous oscillations (5 Hz, 1 cmH2O amplitude, 2 cmH20 peak to peak). Response to the oscillations was analyzed to calculate ∆Xrs and EPAP was adjusted automatically between 4 and 20 cmH2O. A fixed pressure support of 6 cmH2O was delivered. ∆Xrs was measured sitting and supine. Participants with evidence of EFLT (∆Xrs > 2.8) were asked to undergo overnight polysomnography (PSG) and then a sub-group of patients used the ventilator at home for two weeks. EFLT within and between participants was analyzed. EFLT behavior during PSG, the response of the device to dynamically abolish EFLT, as well as the impact of this therapy on sleep quality was studied. Objective ventilator adherence data were used to determine usage after the 2-week in-home use. Additionally, experienced NIV participants qualitatively rated therapy comfort compared to their current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40 years of age; < 80 years of age
2. Ability to provide consent
3. Diagnosis of COPD
4. Must present with EFL via screening of the vector device at 3 cmH2O
5. Have an EPAP to abolish EFL greater or equal to 6cmH2O
6. Must be able to maintain SpO2 greater than 88% at rest and during EPAP Titration
7. Participants who completed the initial study and who would be willing to use the Vector NIV device at home during the night for a 2 week period OR
8. Participants prescribed and currently using a PAP or NIV device at home who meet study inclusion/exclusion criteria of primary protocol

Exclusion Criteria:

1. Any major non COPD uncontrolled disease or condition, such as congestive heart failure, malignancy, liver or renal insufficiency (that requires current evaluation for liver or renal transplantation or dialysis), amyotrophic lateral sclerosis, or severe stroke, or other condition as deemed appropriate by investigator as determined by review of medical history and / or participant reported medical history
2. Suffering from a COPD exacerbation at the time of data collection or in the 30 days prior to data collection
3. Self-reported Pregnancy
4. Employee or family member that is affiliated with Philips Respironics
5. Currently employed by a manufacturer of respiratory products or family member employed by a manufacturer of respiratory products
6. History of bullous emphysema
7. History of pneumothorax
8. Evidence of acute sinusitis or otitis media
9. Hypotension
10. Participants at risk for aspiration of gastric contents
11. Epistaxis
12. Participants in respiratory failure
13. Inability to maintain a patent airway or adequately clear secretions
14. Participants currently using a PAP or NIV device at home with a documented EPAP setting on their current device that is greater than then the mean or final EPAP determined during the therapy session of the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pulmonary Rehabilitation Associates, Youngstown, Ohio
  - Jefferson Associates and Internal Medicine, Clairton, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKenzie J, Nisha P, Cannon-Bailey S, Cain C, Kissel M, Stachel J, Proscyk C, Romano R, Hardy B, Calverley PMA. Overnight variation in tidal expiratory flow limitation in COPD patients and its correction: an observational study. Respir Res. 2021 Dec 23;22(1):319. doi: 10.1186/s12931-021-01913-7. PMID 34949190

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | Auto-titrating EPAP
Started | 42
Completed | 15
Not Completed | 27
Not completed — Screen Failure | 26
Not completed — Withdrawal by Subject | 1
Period: Overnight Polysomnography (PSG)
Arm/Group | Auto-titrating EPAP
Started | 15
Completed | 15
Not Completed | 0
Period: 2 Week Take Home
Arm/Group | Auto-titrating EPAP
Started | 15
Completed | 10
Not Completed | 5
Not completed — Screen Fail | 5

BASELINE CHARACTERISTICS:
Population: All participants that signed a consent form.
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (7.0)
Forced Expiratory Volume in one second / Forced Vital Capacity [Mean (Standard Deviation); unit: percentage] — Population: Historical Spirometry data was collected not all participants had the FEV1/FVC values available.
  percentage
    number analyzed (Participants) | 36
    (all) | 55.2 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Average EPAP During Overnight PSG
Description: The expiratory positive airway pressure (EPAP) is the parameter that is automatically adjusted. The ventilator automatically titrates EPAP to the minimum value able to abolish expiratory flow limitation.
Time Frame: Approximately 8 hours
Population: PSG data was not available for one participant.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 14
cmH2O | 9.5 (5.4)

2. Primary Outcome: Difference Between Mean Inspiratory and Expiratory Reactance During Overnight PSG
Description: The difference between mean inspiratory and expiratory reactance is measured using the forced oscillation technique. The difference between mean inspiratory and expiratory reactance is an index of tidal expiratory flow limitation. Values > 2.8 cmH2O*s/L are indicative of tidal expiratory flow limitation.
Time Frame: Approximately 8 hours
Measure: Mean (Standard Deviation); unit: cmH20/L/s
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 15
cmH20/L/s | 2.7 (5.4)

3. Primary Outcome: Average EPAP for 2 Week Device Take Home Studies
Description: as for outcome 1
Time Frame: Approximately 8 hours nightly use over 14 days
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 10
cm H2O | 6.4 (1.3)

4. Primary Outcome: Difference Between Mean Inspiratory and Expiatory Reactance During 2 Week Device Take Home Studies
Description: The difference between mean inspiratory and expiatory reactance is measured using the forced oscillation technique. The difference between mean inspiratory and expiratory reactance is an index of tidal expiratory flow limitation. Values > 2.8 cmH2O*s/L are indicative of tidal expiratory flow limitation.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cmH20/L/s
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 10
cmH20/L/s | 2.25 (0.9)

5. Secondary Outcome: Sleep Quality
Description: Sleep quality is a key outcome during overnight studies. Nocturnal non-invasive ventilation may affect sleep quality in two ways: 1) it may improve it by reducing sleep-related respiratory problems; 2) it may worsen it if the ventilation mode causes discomfort to the patient. Sleep quality was evaluated by full laboratory polysomnography. Participants after there overnight answered a question of comfort and they answered as 1- being very uncomfortable 2- uncomfortable 3- neutral 4- comfortable 5- very comfortable.
Time Frame: Approximately 8 hours
Population: 2 participants completed a different version of the questionnaire. 1 participant did not morning assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 7
Participants
  Comfortable | 2
  Very Comfortable | 5

6. Secondary Outcome: 2 Week Home Use Device Compliance
Description: Device usage every day, for 14 days based on data downloaded from the device.
Time Frame: Nightly use for 14 days
Measure: Mean (Standard Deviation); unit: hours of therapy per night
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 10
hours of therapy per night | 7.2 (4.3)

7. Secondary Outcome: Therapy Comfort Survey
Description: Prior NIV users rated their comfort with the Forced Oscillation Technique (FOT) therapy over their prior non-invasive ventilation (NIV) therapy. Participants were asked the question "how comfortable did the pressure therapy feel compared to your current device" and they answered the questions on a scale of 0 to 5.
  5-Very Comfortable 4-Comfortable 3-Neutral 2-Uncomfortable
  1-Very Uncomfortable 0-Not applicable
Time Frame: End of 2 weeks device take home study
Population: 2 participants did not complete final assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-titrating EPAP
Number analyzed (Participants) | 8
Participants
  Not Applicable | 4
  Uncomfortable | 1
  Very Comfortable | 3

ADVERSE EVENTS:
Time Frame: Through 2 week take home
Arm/Group | Auto-titrating EPAP
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-titrating EPAP (N=42)
Alcohol detox (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-titrating EPAP (N=42)
Cold (Immune system disorders) | 1 (1)
Acute COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT04725500/Prot_SAP_000.pdf